CLINICAL TRIAL: NCT01095471
Title: A follow-on, Multi-centre, Open-label, Clinical, Phase 4 Trial to Investigate the Persistence of Serotype-specific Antibodies at 40 Months of Age in Children Who Have Received Either the 7-valent or the 13-valent Pneumococcal Conjugate Vaccine at 2, 4 and 12 Months of Age and Assessing the Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine Booster Dose Given at 40 Months of Age
Brief Title: 13 Valent Pneumococcal Conjugate Vaccine - Follow-on Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Bristol (Other); University of Southampton (Other); University of London (Other)
Responsible Party: Professor Andrew Pollard, Chief Investigator, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009/04
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Pneumococcal Disease
Keywords: 7 valent Pneumococcal conjugate vaccine; 13 valent Pneumococcal conjugate vaccine; PCV13; PCV7
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCV13 (Experimental): Initial vaccination with PCV13
  Interventions: Biological: PCV13
- PCV7 (Experimental): Initial intervention with PCV7
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: PCV13 — Immunisation with the 13-valent pneumococcal conjugate vaccine (PCV13) at approximately 40 months of age.
  Other Names: 13-valent pneumococcal conjugate vaccine

SUMMARY:
This is a follow-on, multi-centre, open-label, clinical trial. The purpose of this trial is to investigate the concentrations of serotype-specific antibodies to IgG included in PCV13 in children who have received either the PCV7 or PCV13 primary immunisation at 2, 4 and 12 months of age. We intend to recruit all interested participants who completed the Wyeth-sponsored PCV13 infant trial study (6096A1-007) at selected study sites (i.e. those that recruited the majority of the children in the original study). The study will start in March 2010, at which time the eldest participants in the 6096A1-007 study will be approximately 42 months of age. There will be two visits per participant, 1 month apart from each other. At visit one, all participants will have a blood test and receive a dose of PCV13. At visit 2, all participants will have a blood test and will be offered the remaining pre-school booster vaccinations unless they have already received them.

ELIGIBILITY:
Inclusion Criteria:

1. Participant completed the Wyeth-sponsored PCV13 infant trial study (6096A1-007) at one of the study sites participating in this follow-on study.
2. Aged 39-46 months (inclusive) at time of enrolment.
3. Available for entire study period and whose parent/legal guardian can be reached by telephone.
4. Healthy children as determined by medical history, physical examination, done by a study nurse (and/or study doctor if required, depending on the medical history of the participant and physical assessment), and judgment of the investigator.
5. Parent/legal guardian must be able to complete all relevant study procedures during study participation.

Exclusion Criteria:

1. Has received further doses of pneumococcal vaccination with licensed or investigational pneumococcal vaccine other than those given as part of the Wyeth-sponsored PCV13 infant trial study (6096A1-007).
2. A previous anaphylactic reaction to any vaccine or vaccine-related component.
3. Contraindication to vaccination with pneumococcal conjugate vaccine.
4. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
5. Known or suspected immune deficiency or suppression.
6. History of culture-proven invasive disease caused by S pneumoniae.
7. Major known congenital malformation or serious chronic disorder.
8. Significant neurologic disorder or history of seizures including febrile seizure, or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorder.
9. Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies; eg, synagisB).
10. Participation in another investigational study other than the Wyeth-sponsored PCV13 infant trial study (6096A1-007). Participation in purely observational studies is acceptable.
11. Child who is a direct descendant (child, grandchild) of the study site personnel.

Ages: 39 Months to 46 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of PCV13 booster vaccinations | 1 month
  To assess the proportion of participants, immunised with the 13-valent pneumococcal conjugate vaccine (PCV13) at 2, 4 and 12 months of age, who have IgG concentrations ≥ 0.35mcg/ml for PCV13 serotypes at the time when preschool booster vaccinations are due (at 40 months of age).

SECONDARY OUTCOMES:
To assess IgG concentrations for PCV13 serotypes in children immunised with PCV7 and PCV13 | 1 month
  To assess the proportion of participants, immunised with the 7-valent pneumococcal conjugate vaccine (PCV7) at 2, 4 and 12 months of age, who have IgG concentrations ≥ 0.35mcg/ml for PCV13 serotypes at the time when preschool booster vaccinations are due (at 40 months of age) and comparing these to the proportion of participants achieving this threshold after infant immunisation with PCV 13.
Compare PCV13 serotype-specific IgG geometric mean concentrations, opsonophagocytic activity geometric mean titres & the proportion of participants with PCV13 serotype-specific OPA titres ≥ 1:8 (at 40 months) when immunised in infancy with PCV7 or PCV13. | 1 month
Compare PCV serotype-specific IgG GMCs, OPA GMTs & proportion of participants with IgG concs ≥ 0.35mcg/ml & OPA titres ≥ 1:8 one month after booster dose of PCV13 at 40 months in children previously immunised with PCV7 & PCV13 at 2,4 & 12 months. | 1 month
To determine reactogenicity of the pre-school PCV13 booster in terms of rates of local and systemic reactions following vaccination. | 1 month
Investigate influence of genetic polymorphisms on the above immunological markers following infant immunisation with PCV7/PCV13 & following booster dose of PCV13 at 40 months & on the nature of adverse reactions observed after booster. | 1 month
Measure pneumococcal serotype-specific memory B cells frequencies before & 1 month after PCV13 dose (40 months) in subset previously immunised with PCV7/PCV13 at 2,4 & 12 months (serotype studies to include 4,14,23F (present in PCV7) & 1,3,19A). | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, FRCPCH, PhD, Principal Investigator — University of Oxford, Department of Paediatrics
Locations (4):
- United Kingdom (4):
  - Bristol Children's Vaccine Centre, University of Bristol, Bristol
  - St George's Vaccine Institute, University of London, London
  - Oxford Vaccine Group, Dept Paediatrics, University of Oxford, Oxford
  - Wellcome Trust Clinical Research Facility, University of Southampton, Southampton

REFERENCES:
- [Derived] Truck J, Thompson A, Morales-Aza B, Clutterbuck EA, Voysey M, Clarke E, Snape MD, Kelly DF, Finn A, Pollard AJ. Memory B cell response to a PCV-13 booster in 3.5year old children primed with either PCV-7 or PCV-13. Vaccine. 2017 May 9;35(20):2701-2708. doi: 10.1016/j.vaccine.2017.03.079. Epub 2017 Apr 6. PMID 28392142
- [Derived] Truck J, Snape MD, Tatangeli F, Voysey M, Yu LM, Faust SN, Heath PT, Finn A, Pollard AJ. Pneumococcal serotype-specific antibodies persist through early childhood after infant immunization: follow-up from a randomized controlled trial. PLoS One. 2014 Mar 11;9(3):e91413. doi: 10.1371/journal.pone.0091413. eCollection 2014. PMID 24618837